CLINICAL TRIAL: NCT03296813
Title: TRANSFORM-HF: ToRsemide compArisoN With furoSemide FORManagement of Heart Failure
Acronym: TRANSFORM-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080595; U01HL125511-01A1 (NIH)
Record Dates: First submitted 2017-09-26; First posted 2017-09-28 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: loop diuretic
MeSH Terms: conditions — Heart Failure | interventions — Torsemide; Furosemide

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, unblinded, two-arm, multi-center clinical trial of patients with heart failure who are hospitalized. Patients will be randomized 1:1 to either oral torsemide OR oral furosemide prior to hospital discharge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Torsemide (Active Comparator): Oral dosing of torsemide compared to furosemide will be 1mg:2-4mg.
  Interventions: Drug: Torsemide
- Furosemide (Active Comparator): Oral dosing of torsemide compared to furosemide will be 1mg:2-4mg.
  For patients receiving loop diuretics other than furosemide, conversion to furosemide equivalents will be as follows:
  1 mg oral torsemide = 2-4 mg oral furosemide
  1 mg oral or intravenous bumetanide = 40 mg oral furosemide
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Torsemide — Loop diuretic
  Arms: Torsemide
Drug: Furosemide — Loop diuretic
  Arms: Furosemide

SUMMARY:
TRANSFORM-HF is a large-scale, pragmatic, randomized, unblinded clinical effectiveness study comparing torsemide versus furosemide as treatment for heart failure. Approximately 6,000 patients with heart failure will be enrolled. The primary objective of the TRANSFORM-HF study is to compare the treatment strategy of torsemide versus furosemide on clinical outcomes over 12 months in patients with heart failure who are hospitalized.

DETAILED DESCRIPTION:
* This study will be a randomized, unblinded, two-arm, multi-center clinical trial of patients with heart failure who are hospitalized. Heart failure need not be the reason for hospitalization. Patients will be randomized 1:1 to either oral torsemide OR oral furosemide prior to hospital discharge. Oral dosing of torsemide compared to furosemide will be 1mg:2mg. The specific loop diuretic dose will be at the discretion of the treating physician with the above noted conversion.
* Trial enrollment occurs before hospital discharge, at the discretion of the healthcare provider.
* As appropriate, adherence to the randomized medication will be encouraged during the remainder of hospitalization and will continue post-discharge. Patients will receive follow-up per standard care without any additional study-specific visits.
* Patients will have 30-day, 6-month and 12-month follow-up phone contacts for assessments of vital status, interval hospitalizations, adherence, and quality of life. "Central follow-up" and collection of hospital discharge summaries via IRB-approved mechanisms. Subsets of patients enrolled early in the study have additional phone contacts beyond 12 months, up to 30 months, at six month intervals, to document vital status.

ELIGIBILITY:
Inclusion Criteria:

1. Patient hospitalized (≥ 24 hours or over a change in calendar date) with worsening of chronic heart failure, or new diagnosis of heart failure AND meets one of the following criteria:

   1. Has a left ventricular ejection fraction (EF) ≤40% within 24 months prior to and including index hospitalization by any method (with most recent value used to determine eligibility)
   2. Has an elevated natriuretic peptide level (either NT-pro-B-type natriuretic peptide or B-type natriuretic peptide) during index hospitalization as measured by local laboratory (with most recent value used to determine eligibility)
2. Plan for a daily outpatient oral loop diuretic regimen upon hospital discharge with anticipated need for long-term loop diuretic use
3. ≥ 18 years of age
4. Signed informed consent

Exclusion Criteria:

1. End-stage renal disease requiring renal replacement therapy
2. Inability or unwillingness to comply with the study requirements
3. History of heart transplant or actively listed for heart transplant
4. Implanted left ventricular assist device or implant anticipated <3 months
5. Pregnant or nursing women
6. Malignancy or other non-cardiac condition limiting life expectancy to <12 months
7. Known hypersensitivity to furosemide, torsemide, or related agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2973 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Velazquez, MD, Principal Investigator — Yale University; Robert Mentz, MD, Principal Investigator — Duke University
Locations (60):
- United States (60):
  - Russel Medical Center, Alexander City, Alabama
  - The Heart Center, PC, Huntsville, Alabama
  - University of Arizona, Tucson, Arizona
  - V.A. Greater Los Angeles Healthcare System, Los Angeles, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale, New Haven, Connecticut
  - West Haven VA Medical Center, West Haven, Connecticut
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida - Gainesville, Gainesville, Florida
  - Emory Health Care, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Queens Medical Center, Honolulu, Hawaii
  - Fox Valley Clinical Research Center, Aurora, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Indiana University Health Bloomington Hospital, Bloomington, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University Medical Center, New Orleans, Louisiana
  - Oschner Clinic, New Orleans, Louisiana
  - VA Medical Center/University of Maryland, Baltimore, Maryland
  - Shady Grove Medical Center, Rockville, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Joseph Mercy Health System / Michigan Heart, Ypsilanti, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Lester E. Cox Health Systems, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefore Medical Center - Albert Einstein University Hospital, The Bronx, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Duke (Duke Heart Center), Durham, North Carolina
  - Novant Health Matthews Medical Center, Matthews, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Good Samaritan Hospital, Ephrata, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Jefferson University Hospital, Philadelphia, Pennsylvania
  - Main Line Health System, Wynnewood, Pennsylvania
  - Greenville Hospital System University Medical Center, Greenville, South Carolina
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - Baylor University Medical Center, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - Inova Health Care Services, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Health, Richmond, Virginia
  - Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rao VS, Cox ZL, Ivey-Miranda JB, Neville D, Balkcom N, Moreno-Villagomez J, Ramos-Mastache D, Maulion C, Bellumkonda L, Tang WHW, Collins SP, Velazquez EJ, Mentz RJ, Wilson FP, Turner JM, Wilcox CS, Ellison DH, Fang JC, Testani JM. Mechanistic Differences between Torsemide and Furosemide. J Am Soc Nephrol. 2025 Jan 1;36(1):99-107. doi: 10.1681/ASN.0000000000000481. Epub 2024 Aug 28. PMID 39196651
- [Derived] Kittipibul V, Mentz RJ, Clare RM, Wojdyla DM, Anstrom KJ, Eisenstein EL, Ambrosy AP, Goyal P, Skopicki HA, Ketema F, Kim DY, Desvigne-Nickens P, Pitt B, Velazquez EJ, Greene SJ. On-treatment analysis of torsemide versus furosemide for patients hospitalized for heart failure: A post-hoc analysis of TRANSFORM-HF. Eur J Heart Fail. 2024 Jul;26(7):1518-1523. doi: 10.1002/ejhf.3293. Epub 2024 May 15. PMID 38745502
- [Derived] Kapelios CJ, Greene SJ, Mentz RJ, Ikeaba U, Wojdyla D, Anstrom KJ, Eisenstein EL, Pitt B, Velazquez EJ, Fang JC; TRANSFORM-HF Investigators. Torsemide Versus Furosemide After Discharge in Patients Hospitalized With Heart Failure Across the Spectrum of Ejection Fraction: Findings From TRANSFORM-HF. Circ Heart Fail. 2024 Mar;17(3):e011246. doi: 10.1161/CIRCHEARTFAILURE.123.011246. Epub 2024 Mar 4. PMID 38436075
- [Derived] Greene SJ, Velazquez EJ, Anstrom KJ, Clare RM, DeWald TA, Psotka MA, Ambrosy AP, Stevens GR, Rommel JJ, Alexy T, Ketema F, Kim DY, Desvigne-Nickens P, Pitt B, Eisenstein EL, Mentz RJ; TRANSFORM-HF Investigators. Effect of Torsemide Versus Furosemide on Symptoms and Quality of Life Among Patients Hospitalized for Heart Failure: The TRANSFORM-HF Randomized Clinical Trial. Circulation. 2023 Jul 11;148(2):124-134. doi: 10.1161/CIRCULATIONAHA.123.064842. Epub 2023 May 22. PMID 37212600
- [Derived] Mentz RJ, Anstrom KJ, Eisenstein EL, Sapp S, Greene SJ, Morgan S, Testani JM, Harrington AH, Sachdev V, Ketema F, Kim DY, Desvigne-Nickens P, Pitt B, Velazquez EJ; TRANSFORM-HF Investigators. Effect of Torsemide vs Furosemide After Discharge on All-Cause Mortality in Patients Hospitalized With Heart Failure: The TRANSFORM-HF Randomized Clinical Trial. JAMA. 2023 Jan 17;329(3):214-223. doi: 10.1001/jama.2022.23924. PMID 36648467
- [Derived] Eisenstein EL, Sapp S, Harding T, Harrington A, Velazquez EJ, Mentz RJ, Greene SJ, Sachdev V, Kim DY, Anstrom KJ. Ascertaining Death Events in a Pragmatic Clinical Trial: Insights From the TRANSFORM-HF Trial. J Card Fail. 2022 Oct;28(10):1563-1567. doi: 10.1016/j.cardfail.2022.01.020. Epub 2022 Feb 16. PMID 35181553
- [Derived] Greene SJ, Velazquez EJ, Anstrom KJ, Eisenstein EL, Sapp S, Morgan S, Harding T, Sachdev V, Ketema F, Kim DY, Desvigne-Nickens P, Pitt B, Mentz RJ; TRANSFORM-HF Investigators. Pragmatic Design of Randomized Clinical Trials for Heart Failure: Rationale and Design of the TRANSFORM-HF Trial. JACC Heart Fail. 2021 May;9(5):325-335. doi: 10.1016/j.jchf.2021.01.013. Epub 2021 Mar 10. PMID 33714745
- See also: Related Info — http://dcri.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2973 patients consented. 114 not randomized due to patient decision, PI decision, discharge before randomization occurred, died prior to randomization, or did not meet one or more eligibility criteria.
Groups:
- Furosemide: Oral dosing of torsemide compared to furosemide will be 1mg:2-4mg.
  For patients receiving loop diuretics other than furosemide, conversion to furosemide equivalents will be as follows:
  1 mg oral torsemide = 2-4 mg oral furosemide
  1 mg oral or intravenous bumetanide = 40 mg oral furosemide
  Furosemide: Loop diuretic
Period: Overall Study
Arm/Group | Torsemide | Furosemide
Started | 1431 | 1428
Completed | 1378 | 1368
Not Completed | 53 | 60

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Torsemide | Furosemide | Total
Number analyzed (Participants) | 1431 | 1428 | 2859
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (14) | 65 (14) | 64.5 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 498 | 557 | 1055
  Male | 933 | 871 | 1804
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 75 | 80 | 155
  Not Hispanic or Latino | 1355 | 1345 | 2700
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 3 | 12
  Asian | 37 | 26 | 63
  Native Hawaiian or Other Pacific Islander | 13 | 7 | 20
  Black or African American | 474 | 494 | 968
  White | 831 | 837 | 1668
  More than one race | 65 | 58 | 123
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1431 | 1428 | 2859

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality, as Measured by Follow-up Phone Call or NDI
Description: Death information was obtained from the Call Center through 30 months for patients 1-500, through 24 months for patients 501-1000, through 18 months for patients 1001-1500, and through 12 months for the remaining patients (except those who were randomized < 12 months when the study was stopped by the DSMB). Also death information was obtained through searches of the 2018-2021 National Death Index (NDI) database.
Time Frame: up to 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Furosemide
Number analyzed (Participants) | 1431 | 1428
Participants | 373 | 374
Statistical Analysis 1: Comparison: Torsemide vs Furosemide; To determine whether torsemide is superior to furosemide with respect to all-cause mortality among patients hospitalized for heart failure; Test type: Superiority; p = 0.765, Regression, Cox — P-value not adjusted for multiple comparisons; Hazard Ratio (HR) = 1.022, 95% CI 2-sided [0.885 to 1.180]; P-value from a Cox proportional hazards regression model including the assigned treatment (torsemide vs. furosemide as the reference group) as well as age, sex, baseline ejection fraction (<40%, 41-49%, >50%, unknown), and loop diuretic treatment prior to index hospital admission as covariates

2. Secondary Outcome: All-cause Mortality or All-cause Hospitalization, as Measured by Follow-up Phone Call or NDI (for Death)
Description: The time-to-event analysis of all-cause mortality or all-cause primary re-hospitalization was based on the time from randomization through death or the first primary re-hospitalization through 12 months. Patients who died or whose first all-cause re-hospitalization was after month 12 were censored at month 12. Patients who did not have a re-hospitalization and were alive were censored at the minimum of the time of the last re-hospitalization assessment or month 12.
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Furosemide
Number analyzed (Participants) | 1431 | 1428
Participants | 677 | 704
Statistical Analysis 1: Comparison: Torsemide vs Furosemide; To determine whether torsemide is superior to furosemide with respect to all-cause mortality or first all-cause hospitalization through month 12 among patients hospitalized for heart failure; Test type: Superiority; p = 0.113, Regression, Cox — For secondary analyses, a statistically significant p-value < 0.005 was pre-specified to address the multiple planned analyses and help control the overall type I error rate; Hazard Ratio (HR) = 0.918, 95% CI 2-sided [0.826 to 1.020]; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Total Re-hospitalizations, as Measured by Follow-up Phone Call
Description: Total all-cause primary re-hospitalization was defined as a hospitalization after the index hospitalization through month 12 that met one of the following criteria: 1.) at least a 24-hour stay (or a change in calendar date if the time of admission/discharge is not available) or 2.) reported as an in-patient admission by the patient/proxy with an admission date (complete or month and year) and no discharge date (i.e., length of stay could not be derived). Unit of measurement is the total number of re-hospitalizations for each subject (e.g., if a subject had 3 re-hospitalizations, then the outcome is 3 for the subject).
Time Frame: up to 12 months
Population: Participants who had at least one re-hospitalization.
Measure: Number; unit: re-hospitalizations
Arm/Group | Torsemide | Furosemide
Number analyzed (Participants) | 536 | 577
re-hospitalizations | 940 | 987
Statistical Analysis 1: Comparison: Torsemide vs Furosemide; To determine whether torsemide is superior to furosemide with respect to total all-cause hospitalizations through month 12 among patients hospitalized for heart failure; Test type: Superiority; p = 0.366, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.945, 95% CI 2-sided [0.836 to 1.068]; P-value from a negative binomial regression of the frequency of re-hospitalizations with an offset term of the log of each subject's months to last re-hospitalization assessment through month 12. Re-hospitalizations greater than or equal to 5 were combined and analyzed with re-hospitalizations = 5 (i.e., one category >=5) and for the subjects with >=5 re-hospitalizations, the offset term was the log of the months to the 5th re-hospitalization

4. Secondary Outcome: All-cause Mortality or All-cause Hospitalization, as Measured by Follow-up Phone Call or NDI (for Death)
Description: All-cause mortality or all-cause hospitalization over 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Furosemide
Number analyzed (Participants) | 1431 | 1428
Participants | 149 | 157
Statistical Analysis 1: Comparison: Torsemide vs Furosemide; To determine whether torsemide is superior to furosemide with respect to all-cause mortality or first all-cause hospitalization through day 30 among patients hospitalized for heart failure; Test type: Superiority; p = 0.610, Regression, Cox — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.943, 95% CI 2-sided [0.753 to 1.181]; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Health-related Quality of Life (QOL), as Measured by Follow-up Phone Call
Description: QOL as assessed by the Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS) (range, 0-100 with 100 indicating best health status). The KCCQ was administered prior to randomization (collected by the site) and at Months 1, 6 and 12 (ascertained at the Call Center visits). The outcome is the least square means in Torsemide and Furosemide groups where the difference = Torsemide mean minus Furosemide mean at the monthly assessment.
Time Frame: Baseline, 1 month, 6 months, 12 months
Population: Participants with both baseline and monthly KCCQ-CSS scores available (i.e., change from baseline at the month assessment could be analyzed).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Torsemide | Furosemide
Number analyzed (Participants) | 1431 | 1428
score on a scale
  Baseline to Month 1: number analyzed (Participants) | 981 | 996
  Baseline to Month 1 | 69.52 [67.53 to 71.51] | 68.22 [66.22 to 70.23]
  Baseline to Month 6: number analyzed (Participants) | 800 | 826
  Baseline to Month 6 | 70.61 [68.53 to 72.70] | 71.01 [68.91 to 73.10]
  Baseline to Month 12: number analyzed (Participants) | 665 | 656
  Baseline to Month 12 | 70.00 [67.85 to 72.15] | 69.98 [67.80 to 72.16]
Statistical Analysis 1: Comparison: Torsemide vs Furosemide; To determine whether torsemide improves the QOL at 1 month compared to Furosemide as assessed by the KCCQ among patients hospitalized for heart failure; Test type: Superiority; p = 0.194, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.30, 95% CI 2-sided [-0.66 to 3.26]; Least squares means results from mixed-model repeated measures analysis of the KCCQ score change from baseline with terms for treatment, time (visit) from randomization, treatment x time (visit) interaction as well as the baseline KCCQ score, age, sex, baseline ejection fraction (<40%, 41-49%, >50%, unknown), and loop diuretic treatment prior to index hospital admission as covariates
Statistical Analysis 2: Comparison: Torsemide vs Furosemide; To determine whether torsemide improves the QOL at 6 months compared to Furosemide as assessed by the KCCQ among patients hospitalized for heart failure; Test type: Superiority; p = 0.718, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-2.53 to 1.74]; [other analysis details as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Torsemide vs Furosemide; To determine whether torsemide improves the QOL at 12 months compared to Furosemide as assessed by the KCCQ among patients hospitalized for heart failure; Test type: Superiority; p = 0.987, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-2.26 to 2.30]; [other analysis details as in outcome 5, analysis 1]

6. Secondary Outcome: Symptoms of Depression as Measured by the Patient Health Questionnaire-2 (PHQ-2)
Description: Depression was assessed by the Patient Health Questionnaire-2 (PHQ-2) over 12 months. The PHQ-2 inquires about the frequency of depressed mood and anhedonia (inability to feel pleasure) over the past two weeks. The responses to the questions are scored 0 = Not at all, 1 = Several days, 2 = More than half the days, and 3 = Nearly every day. The PHQ-2 total score is obtained by adding the score for each question. The PHQ-2 total score ranges from 0-6. Reported as the number of patients with a total score <3 versus >=3.
Time Frame: Month 1, month 6, month 12
Population: Participants with data available at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Torsemide | Furosemide
Number analyzed (Participants) | 1431 | 1428
Participants
  Month 1: number analyzed (Participants) | 938 | 963
  Month 1: PHQ-2 score < 3 | 790 | 813
  Month 1: PHQ-2 score > = 3 | 148 | 150
  Month 6: number analyzed (Participants) | 771 | 791
  Month 6: PHQ-2 score < 3 | 658 | 672
  Month 6: PHQ-2 score > = 3 | 113 | 119
  Month 12: number analyzed (Participants) | 628 | 619
  Month 12: PHQ-2 score < 3 | 533 | 537
  Month 12: PHQ-2 score > = 3 | 95 | 82
Statistical Analysis 1: Comparison: Torsemide vs Furosemide; To determine whether torsemide reduces symptoms of depression at 1 month compared to Furosemide as assessed by the PHQ-2 among patients hospitalized for heart failure; Test type: Superiority; p = 0.904, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Torsemide vs Furosemide; To determine whether torsemide reduces symptoms of depression at 6 months compared to Furosemide as assessed by the PHQ-2 among patients hospitalized for heart failure; Test type: Superiority; p = 0.829, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Torsemide vs Furosemide; To determine whether torsemide reduces symptoms of depression at 12 months compared to Furosemide as assessed by the PHQ-2 among patients hospitalized for heart failure; Test type: Superiority; p = 0.342, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality data was collected for up to 30 months
Description: Serious and Other Adverse Event data were not collected.
Arm/Group | Torsemide | Furosemide
All-Cause Mortality (participants affected / at risk) | 373/1431 | 374/1428
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT03296813/Prot_SAP_001.pdf
  • Informed Consent Form (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT03296813/ICF_000.pdf